CLINICAL TRIAL: NCT00591591
Title: Absolute Near-Infrared Brain Oximeter
Brief Title: Brain Oxygenation and Hemodynamics During Sleep in Obstructive Sleep Apnea Sufferers
Acronym: NIRS-OSAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ISS, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Carle Foundation Hospital (Other); University of Illinois at Chicago (Other); University of California, Irvine (Other)
Responsible Party: Antonios Michalos, M.D., M.S./Director of Medical Research, Principal Investigator, ISS, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R44NS040597 (NIH); 2R44NS040597-04 (NIH); GRANT00130523 (Other: NIH NINDS); RNS040597C (Other: NIH NINDS)
Record Dates: First submitted 2007-12-21; First posted 2008-01-11 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; sleep disordered breathing; polysomnography (psg); continuous positive airway pressure (cpap); brain vascular autoregulation; brain tissue oxygenation; near-infrared spectroscopy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OSA (Experimental): Persons with suspected obstructive sleep apnea (OSA) undergoning overnight sleep evaluation
  Interventions: Device: OxiplexTS
- Controls (No Intervention): Healthy controls

INTERVENTIONS:
Device: OxiplexTS — OxiplexTS is a Frequency Domain Near-Infrared Tissue oximeter which provides absolute values of tissue oxygenation in real time. It also provides physiological quantities of oxy, deoxy and total hemoglobin concentration, which form the basis for the functional measurement of brain hemodynamics. Both the control and OSA groups will undergo standard overnight sleep study (PSG). In addition to the standard PSG, with or without Continuous Positive Airway Pressure (CPAP), we will add the OxiplexTS, allowing us to assess brain oxygenation and hemodynamics during sleep. The hemodynamic patterns of the healthy controls will be compared to the OSA sufferers. Participants with OSA who undergo PSG/CPAP will be also tested with the OxiplexTS. Their PSGs and PSG/CPAP data will be compared.
  Arms: OSA

SUMMARY:
The goal of this trial is to assess the performance of the OxiplexTS-an absolute near-infrared oximeter-as an instrument to measure brain oxygenation and hemodynamics in sleep medicine as well as in the broader field of cardiovascular/cerebrovascular diagnostics.

DETAILED DESCRIPTION:
Frequency domain near-infrared spectroscopy (NIRS) offers the advantage of performing safe, non-invasive, transcranial, quantitative measurements of brain oxygenation and hemodynamics in real-time. These characteristics make NIRS the ideal tool to study physiological and pathological processes of the brain, in settings ranging from research and diagnostic laboratories to intensive care units and operating rooms.

Scientists recently developed the first commercially available absolute near-infrared oximeter, called OxiplexTS. This portable device will be used to study brain vascular autoregulatory responses (such as responses to hypoxia and hypercapnia) in persons with obstructive sleep apnea (OSA). These responses to allow for the assessment of brain vascular health. The OxiplexTS device will be beneficial in identifying persons at risk for cerebrovascular disease. Polysomnography (PSG), which is currently used to assess sleep disorders, gives important information on the function of different systems, however, it does not provide information on brain oxygenation and hemodynamics during sleep. The assessment of these factors, via NIRS, in persons with OSA is crucial because of the high prevalence of the disorder and the significant cardio/cerebrovascular health risk it represents.

The specific aim of this trial is to make OxiplexTS a clinically usable instrument, especially for research and clinical diagnosis and monitoring of sleep disorders. An additional goal is to determine the usefulness of this instrument for providing measurements in various clinical situations including intensive care management or prolonged surgical procedures, such as cardiothoracic surgery that require critical information of brain oxygenation and hemodynamics. This trial emerges from previous phase I and phase II studies which determined the feasibility of using OxiplexTS to assess brain vascular autoregulatory responses to hypoxic stimuli.

Approximately 300 participants will be recruited from a pool of healthy individuals, individuals with OSA, and volunteers undergoing overnight diagnostic or therapeutic PSG for suspected OSA.

Participants will be divided into two groups: healthy controls and persons with OSA. Both groups will undergo standard overnight sleep study or PSG. In addition to the standard PSG (with or without Continuous Positive Airway Pressure (CPAP)), the study researchers will add the OxiplexTS-allowing them to assess brain oxygenation and hemodynamics during sleep. The hemodynamic patterns of the healthy controls will be compared to those of persons with OSA. Participants with OSA who undergo PSG/CPAP will be tested with the OxiplexTS, as well. Their PSG and PSG/CPAP data will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (controls)
* Individuals undergoing overnight polysomnography foe suspected obstructive sleep apnea

Exclusion Criteria:

* Documented severe cardiovascular disease.
* Documented cerebrovascular disease
* Documented cardiopulmonary disease
* Pregnancy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Michalos, M.D., M.S., Principal Investigator — ISS, Inc.
Locations (4):
- United States (4):
  - University of California-Irvine Sleep Disorders Center, 101 The City Drive South, Bldg. 22C, 2nd Floor, Rt. 23, Orange, California
  - Stanford Sleep Disorders Clinic, Psychiatry Building, 401 Quarry Road, Stanford, California
  - Center of Sleep and Ventilatory Disorders, University of Illinois Medical Center at Chicago, 2200 W Harrison, Chicago, Illinois
  - Carle Regional Sleep Disorders Center, Carle Foundation Hospital, 611 West Park Street, Urbana, Illinois

REFERENCES:
- [Background] Safonova LP, Michalos A , Wolf U, Wolf M, Mantulin WW, Hueber DM and Gratton E. Diminished cerebral circulatory autoregulation in obstructive sleep apnea investigated by near-infrared spectroscopy. Sleep Research on-line 2003; 5(4): 123-132, 2003.
- [Background] Safonova LP, Michalos A, Wolf U, Wolf M, Hueber DM, Choi JH, Gupta R, Polzonetti C, Mantulin WW, Gratton E. Age-correlated changes in cerebral hemodynamics assessed by near-infrared spectroscopy. Arch Gerontol Geriatr. 2004 Nov-Dec;39(3):207-25. doi: 10.1016/j.archger.2004.03.007. PMID 15381340
- [Background] Olopade CO, Mensah E, Gupta R, Huo D, Picchietti DL, Gratton E, Michalos A. Noninvasive determination of brain tissue oxygenation during sleep in obstructive sleep apnea: a near-infrared spectroscopic approach. Sleep. 2007 Dec;30(12):1747-55. doi: 10.1093/sleep/30.12.1747. PMID 18246984
- See also: company website — http://www.iss.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: OSAS sufferers and Controls have been recruited an tested at:
  1. Center of Sleep Disorders of the University of Illinois at Chicago.
  2. Regional Sleep Disorders Center at Carle Foundation Hospital (Urbana,IL).
  3. University of California-Irvine Medical Center-Center for Sleep Disorders (UCIMC)
  4. Stanford University -Sleep Disorders Clinic
Groups:
- Obsructive Sleep Apnea Sufferers: Patients undergoing sleep evaluation for suspected obstructive sleep apnea syndrome
Period: Overall Study
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Started | 176 | 133
Completed | 165 | 94
Not Completed | 11 | 39
Not completed — Withdrawal by Subject | 1 | 37
Not completed — Lack of Efficacy | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers | Total
Number analyzed (Participants) | 176 | 133 | 309
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 176 | 133 | 309
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.9 (10.15) | 41.7 (8.9) | 38.3 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 86 | 197
  Male | 65 | 47 | 112
Region of Enrollment [Number; unit: participants]
  United States | 176 | 133 | 309

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Oxygen Saturation in the Brain During Sleep
Time Frame: 6 hours of sleep
Population: Absolute Brain Oximetry: Quantitative Hemodynamic Responses of Brain During Sleep, in Healthy & OSA Subjects.
Measure: Mean (Standard Deviation); unit: Percentage of brain oxygen saturation
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Number analyzed (Participants) | 176 | 133
Percentage of brain oxygen saturation | 53.462 (8.825) | 53.13 (11.24)

2. Primary Outcome: Oxyhemoglobin Concentration in the Brain During Sleep
Time Frame: 6 hours of sleep
Population: Absolute Brain Oximetry: Quantitative Hemodynamic Responses of Brain During Sleep, in Healthy & OSA Subjects.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Number analyzed (Participants) | 176 | 133
µM | 18.82 (7.81) | 18.36 (7.96)

3. Primary Outcome: Total Hemoglobin Concentration in the Brain During Sleep
Time Frame: 6 hours of sleep
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Number analyzed (Participants) | 176 | 133
µM | 34.38 (11.72) | 33.71 (11.22)

4. Primary Outcome: Deoxy-Hemoglobin Concentration in the Brain During Sleep
Time Frame: 6 hours of sleep
Population: Absolute Brain Oximetry: Quantitative Hemodynamic Responses of Brain During Sleep, in Healthy & OSA Subjects.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Number analyzed (Participants) | 176 | 133
µM | 15.82 (6.73) | 15.41 (4.71)

5. Secondary Outcome: Apnea Hypopnea Index (AHI is the Index of Severity That Combines Apneas and Hypopneas) Determined During the Routine Sleep Study
Time Frame: 6 hours of sleep
Measure: Mean (Standard Deviation); unit: Number of apnea/hypopnea per sleep hour
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Number analyzed (Participants) | 176 | 133
Number of apnea/hypopnea per sleep hour | 1.78 (2.41) | 42.4 (32.6)

ADVERSE EVENTS:
Arm/Group | Controls | Obsructive Sleep Apnea Sufferers
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/133
Other Adverse Events (participants affected / at risk) | 0/176 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No